CLINICAL TRIAL: NCT01964508
Title: The Use of a microRNA Panel to Identify Thyroid Malignancy in FNA Leftover Cells and the Effect of These microRNAs on Target Genes.
Brief Title: microRNA in Thyroid Cancer
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: HM0003-HMO-CTIL
Record Dates: First submitted 2013-10-14; First posted 2013-10-17 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2013-10

CONDITIONS: FNA; microRNA; Thyroid Cancer; Thyroid Nodule
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Nodule | interventions — Biopsy, Fine-Needle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — FNA samples, CDNA, RNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Thyroid nodule: Patients with thyroid nodules undergoing FNA.
  Interventions: Other: Fine needle aspiration

INTERVENTIONS:
Other: Fine needle aspiration

SUMMARY:
Thyroid cancer is the most common endocrine malignancy and its incidence is rapidly increasing. Palpable thyroid nodules are very common, affecting up to 5% of the general population. Nevertheless, only 5% of the thyroid nodules harbor malignancy, hence the obvious need to accurately characterise these nodules. Ultrasound guided fine needle aspiration biopsy (FNAB) is the most important tool in assessing the nature of thyroid nodules, however, in up to 30% of the biopsies the results are indeterminate. In this proposal, the investigators hypothesize that leftover cells in the FNAB needle may be utilized for molecular analysis with an established microRNA panel and distinguish between malignant and benign lesions. Despite established studies on the diagnostic utility of microRNAs in thyroid nodules, the effect of microRNAs on specific target genes involved in thyroid cancer is poorly studied. In this proposal the investigators hypothesize that the microRNAs identified in our panel will affect intracellular pathways by regulating target genes that are involved in thyroid tumorigenesis. The investigators present preliminary data that confirms that microRNA panel may identify malignancy in thyroid nodules. In aim 1 the investigators will identify the expression profile of miRNAs in the different thyroid cancers. the investigators will statistically quantify the threshold of miRNA dysregulation for malignancy on a large number of tumor and benign samples. This will serve as matrix for defining malignancy on the FNAB samples. In aim 2 the investigators will establish a reliable reproducible method to extract RNA from cells left over in FNAB samples. the investigators' preliminary data support the feasibility of the method and it has not been described previously. This will be the first study that will compare cytology results and microRNA panel analysis on the very same FNAB cells. It will mimic the exact clinical scenario that such microRNA panel can be utilized in the future. Finally, in aim 3 the investigators will characterize the effect of microRNAs on target genes expression. the investigators will identify possible target genes from bioinformatics databases and will perform quantitative measurement of mRNA level of target gene by real time PCR and immunohistochemistry. These studies will hopefully support the utility of microRNAs as a diagnostic tool to accurately identify malignancy in thyroid FNAB leftover cells and point out possible target genes for future therapeutic approaches. This could impact many patients, as thyroid cancer is the 5th most common cancer in women, and the most rapidly growing malignancy in both men and women.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing thyroid nodule biopsy; patients signing informed consent

Exclusion Criteria:

* Patients that cannot sign an informed consent form.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing FNA
Sampling Method: Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2013-09-12 (Actual); Primary Completion 2015-12-30 (Actual); Study Completion 2015-12-30 (Actual)

PRIMARY OUTCOMES:
microRNA expression in thyroid cancer | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel